CLINICAL TRIAL: NCT06271993
Title: Skin Prick Test (SPT) for Skin Sensitization (Contact Allergy) of Test Product ColActive Plus Collagen Matrix Dressing
Brief Title: SPT for Sensitization of Collagen Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Covalon Technologies Inc. (Industry)
Collaborators: ALS Beauty and Personal Care (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-233
Record Dates: First submitted 2024-02-15; First posted 2024-02-22 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Allergy Skin; Allergic Skin Reaction

STUDY DESIGN:
Intervention Model Description: This will be a single center, with no randomization or blinding, study design in 20 healthy adult subjects, age 18-70 years. Based on prior experience approximately 30 subjects will be enrolled to ensure 20 subjects complete the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Collagen wound dressing with positive and negative controls (Other): Application of test dressing, histamine, and saline with glycerin to volar forearm skin
  Interventions: Device: ColActivePlus Collagen Matrix Dressing

INTERVENTIONS:
Device: ColActivePlus Collagen Matrix Dressing — The test product, positive control and negative control will be applied directly to the volar forearm skin of the subject. The sites will be a minimum of 2cm from each other to minimize cross contamination.

SUMMARY:
The goal of this clinical trial is to determine the sensitization (contact allergy) potential of the test product ColActive Plus Collagen Matrix Dressing after a skin prick test on the skin of healthy human subjects. The main question it aims to answer is:

• Does the product induce any sensitization (contact allergy) after a skin prick using a UniTest PC (pain control) device in healthy human subjects? Participants will have the test product and both positive and negative controls applied, and skin response will be evaluated by an allergist at 15 minutes, 6 hours, and 24-48 hours post-application to see if sensitization occurs.

DETAILED DESCRIPTION:
This will be a single center, with no randomization or blinding, study design in 30 healthy adult subjects, age 18-70 years. Based on prior experience approximately 30 subjects will be enrolled to ensure 20 subjects complete the study.

Skin response to the test product and both positive and negative controls will be evaluated and measured by an allergist. If the measured diameter is ≥3mm in response to the test product with expected reactions to both the positive and negative controls, the site will be considered a positive allergen.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70
* Sex: Male & Female
* Fitzpatrick: I-V, minimum 10% of panel Fitzpatrick V.
* Individuals who will be able to read, understand and give an informed consent relating to the study they are participating in.
* Individuals who will be free of any dermatological or systemic disorder, which in the Investigator's opinion, could interfere with the study results.
* Individuals who will be in general good health and who will complete a preliminary medical history form mandated by the testing facility.
* Individuals who will be able to and agree to cooperate with the Investigator and clinical staff.
* Individuals who will agree to have test products applied in accordance with the protocol and are able to complete the full course of the study.
* Individuals who have not participated in a similar study in the past 30 days.
* Individuals who agree to refrain from sun tanning/bathing and prolonged exposure to sunlight (outdoors).
* Individuals who are willing to refrain from wetting, wiping, cleanse, and covering the test sites (volar surface of the forearms) between the baseline and up to 48-hour time points.
* Female volunteers who are willing to undergo a urine pregnancy test.
* Individuals willing to refrain from vitamin C (Emergen-C), orange juice and vitamin water for the study duration and two days prior to the SPT test.

Exclusion Criteria:

* Individuals who are currently taking any medications (topical or systemic) that may mask or interfere with the test results (specifically, corticosteroids, topical and/or systemic [except nasal steroids], non steroidal anti-inflammatory drugs [e.g. ibuprofen, Advil, Motrin, aspirin > 325mg/day], antihistamines, and topical/oral immunosuppressive medications).
* Individuals who have a history of any acute or chronic disease that might interfere with or increase the risk on study participation. (e.g., systemic lupus erythematosus, rheumatoid arthritis, HIV positive).
* Individuals who are diagnosed with chronic skin allergies (atopic dermatitis/eczema) or recently treated skin cancer within the last 12 months.
* Individuals who have damaged skin in close proximity to test sites (e.g., sunburn, uneven skin pigmentation, tattoos, scars, excessive hair, active acne papules or other disfigurations).
* Individuals who control their diabetes using insulin.
* Individuals with any history, which in the Investigator's opinion, indicates the potential for harm to the subject or places the validity of the study in jeopardy.
* Female volunteers who indicate that they are pregnant or are planning to become pregnant or nursing.
* Individuals with a known history of hypersensitivity to any cosmetics, personal care products, fragrances, and/or adhesives.
* Individuals that have a history of dermatographism.
* Individuals have a history of frequent skin irritation.
* Employees of ALS.
* Individuals with a known fish allergy.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-02-08 (Actual); Primary Completion 2024-02-16 (Actual); Study Completion 2024-02-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan DeSantis, MHI, BS, Principal Investigator — ALS
Locations (1):
- ALS Beauty and Personal Care, Torrance, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Skin sites
Groups:
- Collagen Wound Dressing: Application of test dressing to volar forearm skin
  One test dressing will be applied directly to the volar forearm skin of the subject. The site will be a minimum of 2cm from the positive and negative controls to minimize cross contamination.
- Postitive Control: Application of histamine to volar forearm skin
  One positive control will be applied directly to the volar forearm skin of the subject. The site will be a minimum of 2cm from the test and negative control to minimize cross contamination.
- Negative Control: Application of saline with glycerin to volar forearm skin
  One negative control will be applied directly to the volar forearm skin of the subject. The site will be a minimum of 2cm from the test and positive control to minimize cross contamination.
Period: Overall Study
Arm/Group | Collagen Wound Dressing | Postitive Control | Negative Control
Started | 27; 27 Skin sites | 27; 27 Skin sites | 27; 27 Skin sites
Completed | 22; 22 Skin sites | 22; 22 Skin sites | 22; 22 Skin sites
Not Completed | 5; 5 Skin sites | 5; 5 Skin sites | 5; 5 Skin sites
Not completed — Not reactive to histamine | 5 | 5 | 5

BASELINE CHARACTERISTICS:
Arm/Group | Collagen Wound Dressing With Positive and Negative Controls
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: African American | 4
  Race: Asian | 4
  Race: Caucasian | 4
  Race: Hispanic | 8
  Race: Other | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22
Fitzpatrick Skin Type [Count of Participants; unit: Participants]
  I - always burn, does not tan | 2
  II - burn easily, tan slightly | 6
  III - burn moderately, tan progressively | 4
  IV - burn a little, always tan | 6
  V - rarely burn, tan intensely | 4
  VI - never burn, tan very intensely | 0

OUTCOME MEASURES:

1. Primary Outcome: Wheal Measurement
Description: The wheal of each test site will be measured in millimeters. A larger wheal (≥3 mm) is associated with sensitization.
Time Frame: 15-20 minutes following application
Measure: Mean (Full Range); unit: mm
Units Other Than Participants: Skin sites
Groups:
- Collagen Wound Dressing: Application of test dressing to volar forearm skin
  The test product, positive control and negative control will be applied directly to the volar forearm skin of the subject. The sites will be a minimum of 2cm from each other to minimize cross contamination.
- Positive Controls: Application of histamine to volar forearm skin
  The test product, positive control and negative control will be applied directly to the volar forearm skin of the subject. The sites will be a minimum of 2cm from each other to minimize cross contamination.
- Negative Controls: Application of saline with glycerin to volar forearm skin
  The test product, positive control and negative control will be applied directly to the volar forearm skin of the subject. The sites will be a minimum of 2cm from each other to minimize cross contamination.
Arm/Group | Collagen Wound Dressing | Positive Controls | Negative Controls
Number analyzed (Participants) | 22 | 22 | 22
Number analyzed (Skin sites) | 22 | 22 | 22
mm | 0 [0 to 0] | 7.91 [4 to 14] | 0.32 [0 to 4]

2. Primary Outcome: Wheal Measurement
Description: The wheal of each test site will be measured in millimeters. A larger wheal (≥3 mm) is associated with sensitization.
Time Frame: 6 hours (+/-30 minutes)
Measure: Mean (Full Range); unit: mm
Units Other Than Participants: Skin sites
Arm/Group | Collagen Wound Dressing | Positive Controls | Negative Controls
Number analyzed (Participants) | 22 | 22 | 22
Number analyzed (Skin sites) | 22 | 22 | 22
mm | 0 [0 to 0] | 0.27 [0 to 4] | 0.14 [0 to 3]

3. Primary Outcome: Wheal Measurement
Description: The wheal of each test site will be measured in millimeters. A larger wheal (≥3 mm) is associated with sensitization.
Time Frame: 24-48 hours
Measure: Mean (Full Range); unit: mm
Units Other Than Participants: Skin sites
Arm/Group | Collagen Wound Dressing | Positive Controls | Negative Controls
Number analyzed (Participants) | 22 | 22 | 22
Number analyzed (Skin sites) | 22 | 22 | 22
mm | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

ADVERSE EVENTS:
Time Frame: 2 days
Description: Adverse events are graded on a scale of severity (mild, moderate, severe, or life-threatening) and on a scale of relationship to the product (unknown, unrelated, unlikely, possible, probable, or definite). All AEs will be reported to the Sponsor within five business days. All AEs will be followed up until resolved, stabilized, the subject is lost to follow-up or the event is otherwise explained. All serious adverse events will be reported to the Sponsor within 24 hours.
Arm/Group | Collagen Wound Dressing With Positive and Negative Controls
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-29): https://cdn.clinicaltrials.gov/large-docs/93/NCT06271993/Prot_SAP_000.pdf